CLINICAL TRIAL: NCT07214181
Title: Topical Amitriptyline 1% Gel for the Treatment of Burning Mouth Syndrome
Acronym: TOP-AMI → TOPi
Status: Completed | Type: Observational
Sponsor: Universidad de Murcia (Other)
Responsible Party: Principal Investigator, Pia Lopez Jornet, MD, DDS,PhD, Universidad de Murcia
Other Study IDs: C.I. EST: 53/25
Record Dates: First submitted 2025-10-02; First posted 2025-10-09 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: Burning Mouth Syndrome; Stomatodynia
Keywords: pain , Amitriptyline ; treatment
MeSH Terms: conditions — Burning Mouth Syndrome; Stomatodynia; Pain | interventions — Amitriptyline; Gels

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 4 Weeks
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- This retrospective cohort includes patients diagnosed with burning mouth syndrome (BMS: Patients diagnosed with burning mouth syndrome (BMS) according to international diagnostic criteria who received treatment with topical amitriptyline 1% gel. Patients applied the gel intraorally for several weeks as part of routine clinical care. Data collected from medical records included pain intensity (0-10 numerical rating scale) before and after treatment, patient global impression of improvement, and reported adverse events. The cohort reflects real-world use of topical amitriptyline gel for BMS.
  Interventions: Drug: Topical amitriptyline 1% gel

INTERVENTIONS:
Drug: Topical amitriptyline 1% gel — Patients diagnosed with burning mouth syndrome received topical amitriptyline 1% gel applied intraorally. The gel was instructed to be placed on the oral mucosa (tongue and/or other symptomatic areas) two times per day for several weeks, without swallowing. Treatment was provided as part of routine clinical care. This retrospective study collected data on pain intensity, patient global impression of improvement, and adverse events to evaluate the real-world effectiveness and tolerability of this topical formulation.

SUMMARY:
Burning mouth syndrome (BMS) is a chronic oral pain condition that causes a persistent burning or stinging sensation in the mouth, often without visible changes in the tissues. It mostly affects women in midlife and older age and can greatly reduce quality of life.

This study reviewed the medical records of patients with BMS who were treated with a topical 1% amitriptyline gel. The aim was to evaluate whether this gel could reduce pain and to record any side effects.

Patients applied the gel inside the mouth for several weeks. Pain intensity was measured using a 0-10 scale before and after treatment. We also collected information about patients' overall impression of improvement and any reported adverse events.

By analyzing these retrospective data, we hope to provide real-world evidence on the effectiveness and safety of topical amitriptyline gel as a potential treatment option for patients with burning mouth syndrome.

DETAILED DESCRIPTION:
Burning mouth syndrome (BMS) is a chronic oral pain condition that causes a persistent burning or stinging sensation in the mouth, often without visible changes in the tissues. It mostly affects women in midlife and older age and can greatly reduce quality of life.

This study reviewed the medical records of patients with BMS who were treated with a topical 1% amitriptyline gel. The aim was to evaluate whether this gel could reduce pain and to record any side effects.

Patients applied the gel inside the mouth for several weeks. Pain intensity was measured using a 0-10 scale before and after treatment. We also collected information about patients' overall impression of improvement and any reported adverse events.

By analyzing these retrospective data, we hope to provide real-world evidence on the effectiveness and safety of topical amitriptyline gel as a potential treatment option for patients with burning mouth syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients diagnosed with burning mouth syndrome (BMS) according to international diagnostic criteria (ICHD-3 and ICOP).

Symptoms recurring daily for >50% of the day for at least 3 months.

Pain intensity ≥4 on a 0-10 numerical rating scale (NRS) at baseline.

Normal appearance of the oral mucosa and normal intraoral clinical examination.

Received topical amitriptyline 1% gel as part of routine care.

Exclusion Criteria:

* Missing or incomplete medical records.Use of other concomitant topical treatments on the oral mucosa during the study period.
* Change in systemic pain medication while using topical amitriptyline gel.
* Presence of local conditions and sytemic that could cause burning mouth symptoms (e.g., candidiasis, lichen planus, allergies, ).

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: This retrospective study included adult patients diagnosed with burning mouth syndrome (BMS) according to international diagnostic criteria. All patients received topical amitriptyline 1% gel as part of routine clinical care and had complete medical records with baseline and 4-week follow-up data available for analysis.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2024-01-02 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2025-05-30 (Actual)

PRIMARY OUTCOMES:
Title: Change in mean pain intensity (NRS 0-10) | Baseline to 4 weeks after treatment initiation
  Description: Pain intensity measured using a numerical rating scale (0 = no pain, 10 = worst possible pain). Mean daily score calculated from patient records at baseline (before treatment) and after 4 weeks of topical amitriptyline gel.

SECONDARY OUTCOMES:
Patient Global Impression of Improvement (PGI-I) | Time Frame: At 4 weeks
  Description: Patient-reported overall improvement, categorized as "very much better," "much better," "a little better," "no change," or "worse."

CONTACTS AND LOCATIONS:
Locations (1):
- Clinica Odontologica Universitaria, Murcia, Murcia, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Kung CP, Sil BC, Zhang Y, Hadgraft J, Lane ME, Patel B, McCulloch R. Dermal delivery of amitriptyline for topical analgesia. Drug Deliv Transl Res. 2022 Apr;12(4):805-815. doi: 10.1007/s13346-021-00982-x. Epub 2021 Apr 22. PMID 33886076
- [Result] Lebel A, Da Silva Vieira D, Boucher Y. Topical amitriptyline in burning mouth syndrome: A retrospective real-world evidence study. Headache. 2024 Oct;64(9):1167-1173. doi: 10.1111/head.14818. Epub 2024 Aug 23. PMID 39177013